CLINICAL TRIAL: NCT05530941
Title: Evaluation of an Online Suicide Prevention Campaign Aimed at Men to Promote Help-seeking and Peer Support
Brief Title: Online Suicide Prevention Campaign Aimed at Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EC/BC-11283
Record Dates: First submitted 2022-05-31; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-01

CONDITIONS: Help-Seeking Behavior; Suicide
MeSH Terms: conditions — Help-Seeking Behavior; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Participants in this group (all participants) were asked to complete a questionnaire and then received access to the online prevention campaign during three days, after which they were asked to complete another questionnaire.
  Interventions: Behavioral: Online suicide prevention campaign

INTERVENTIONS:
Behavioral: Online suicide prevention campaign — The online prevention campaign consists of two campaign videos, a website with information about suicide prevention and mental health tailored to men, and testimonials of men who struggled with their mental health.

SUMMARY:
This study aims to examine whether the online suicide prevention campaign for men could increase openness about emotions and help-seeking behavior, and decrease hopelessness and adherence to traditional gender norms concerning self-reliance among men. The effectiveness of the campaign will be evaluated in adult men using a pre-post questionnaire study design.

ELIGIBILITY:
Inclusion Criteria:

* Gender identity: male
* ≥ 18 years old
* Have access to internet and a computer/tablet/smartphone
* Speak Dutch

Exclusion Criteria:

* Gender identity: female or other
* < 18 years old
* No acces to internet and a computer/tablet/smartphone
* Non-Dutch speaking

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Change in self-reliance: self-reliance factor of the Conformity to Masculine Norms Inventory (CMNI) | Change from Baseline (before intervention) to post-test (after three days of access to the campaign)
  The CMNI is a 22 item scale to measure adherence to traditional Western masculine norms and values across 11 domains. The self-reliance scale consists of 5 items measured on a 4-point Likert scale (1= strongly disagree to 4= strongly agree).
Change in Help-seeking behaviour: General Help-Seeking Questionnaire (GHSQ) | Change from Baseline (before intervention) to post-test (after three days of access to the campaign)
  The GHSQ measures two aspects of help-seeking, namely when facing personal or emotional problems and when facing suicidal ideation. For each aspect participants indicate how likely (1= extremely unlikely, 7= extremely likely) it is that they would seek help from different kind of sources (10 types).
Change in Openness about emotions: scales "Communication and Expression of Emotions" and "Normative Restrictions of Affectivity" of the Dimensions of Openness to Emotions (DOE) | Change from Baseline (before intervention) to post-test (after three days of access to the campaign)
  The Dimensions of Openness to Emotions is a 36 item questionnaire measuring emotional openness.
  The "Communication and Expression of Emotions" and "Normative Restrictions of Affectivity" consist of, respectively, 7 and 5 items to be scored on a 5-point Likert scale (0=not at all, 4= completely)
Change in Hopelessness: Beck Hopelessness Scale (BHS), 4-item version | Change from Baseline (before intervention) to post-test (after three days of access to the campaign)
  A 4-item self-report questionnaire to measure hopelessness in adolescents and adults. Each item is rated as 'true' (score = 1) or 'false' (score = 0) for them over the past week, resulting in a total score ranging from 0 to 4, with higher scores indicating higher levels of hopelessness.

OTHER OUTCOMES:
General distress: Kessler 10 | Baseline (before intervention)
  A 10-item questionnaire measuring distress. Each item is scored on a 5-point Likert (1=never, 5=always)
Suicidal ideation and behaviour: Suicidal ideation Attributes Scale & two general questions | Baseline (before intervention)
  A 5-item questionnaire to measure presence of suicidal thoughts and the severity of these thoughts. Each item is scored on a 11-point Likert scale.
  Participants were asked whether they ever had had suicidal thoughts (if yes, in the last 12 months?) and whether they ever (if yes, in the last 12 months?) had attempted suicide.
Campaign evaluation | post-test (after three days of access to the campaign)
  14 evaluative statements about the general campaign and specific aspects of the campaign to be rated on a 5-point Likert scale (Totally disagree, disagree, neutral, agree, totally disagree). Additionally three open questions where participants can give feedback about what they liked/did not like/ general comments.

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, Phd, Principal Investigator — University Ghent
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No